CLINICAL TRIAL: NCT01361906
Title: Effects of Sensomotoric Training on Neck/Scapular Pain in People With Visual Disability
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre for Rehabilitation Research, Örebro (Other Government)
Collaborators: Örebro County Council (Other Government); University of Gavle (Other)
Responsible Party: Principal Investigator, Lars-Olov Lundqvist, Research Director, Centre for Rehabilitation Research, Örebro
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REHSAM/11
Record Dates: First submitted 2011-05-25; First posted 2011-05-27 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: Neck/Scapular Pain
Keywords: Musculoskeletal and Neural Physiological Phenomena; Postural Balance; Eye/hand coordination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Untreated control (No Intervention): Untreated control
- Sensomotoric training (Experimental): Treatment with Sensomotoric training
  Interventions: Behavioral: Sensomotoric training

INTERVENTIONS:
Behavioral: Sensomotoric training — The intervention will be given once a week (2h per occasion) for twelve weeks.
  Each occasion is planned to have the following structure:
  10 min initial conversation about how participants are feeling today and how it felt after the last time.
  70 min guided sensory motor learning. 10 min final talks, reflections on how it felt today.
  Arms: Sensomotoric training

SUMMARY:
The purpose of this study is to determine whether sensomotoric training can reduce neck/scapular pain in people with visual disability.

DETAILED DESCRIPTION:
People with prolonged musculoskeletal disorders have impaired quality of life, physical function, work conditions and work ability and consume substantial public resources. An often overlooked fact in this context is the relationship between musculoskeletal disorders and the importance of a normally functioning visual system. People who have a visual impairment in adulthood often experience reduced health and life satisfaction. Many people lose their faith in order to continue with the activities previously carried out as to cope with their life, their work, and in some cases,personal care. Rehabilitative efforts to reduce the negative effects often involve the prescription of various visual aids which, in turn, often leads to unfavourable ergonomic and static postures with further increased risk of musculoskeletal problems. A prevention of such disorders is likely to allow them to continue their work, which is important from both an individual and a society perspective. The overall objective of the project is to evaluate the effects of an intervention program and develop a theoretical model for the relationship between near work, eye disorders and musculoskeletal disorders. The intervention is to be evaluated in a randomized trial on people with impaired vision and pain in the neck and scapular area. An intervention based on development and adaptation of an established physiotherapy practice in order to increase body awareness, body control and movement patterns will be evaluated. The effects of the intervention will be measured by a variety of outcome measures derived from WHO's ICF-model. An innovative solution for establishing proprioception and eye-hand coordination in everyday activities, the Clinical Kinematic Assessment Tool, will be used.

ELIGIBILITY:
Inclusion Criteria:

* visual disability
* age 18 to 67 years old
* pain in neck/scapular area
* living in Örebro county

Exclusion Criteria:

* deafness
* musculoskeletal disease (such as Multiple sclerosis, etc)

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2010-09; Primary Completion 2012-01 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in neck/scapular pain at 12 month | baseline and 12 months
  Physiotherapeut palpation of left and right M.Trapezius, M.Occiput, and M.Levator scapulae. Patient rate degree of pain on 100 mm VAS.

SECONDARY OUTCOMES:
Change from Baseline in sick leave at 12 month | baseline and 12 month
  Patient self reported sick leave and sickleave registered at persons employer (if any) and/or at the Swedish Social Insurance Agency

CONTACTS AND LOCATIONS:
Overall Officials: Lars-Olov Lundqvist, Associate Professor, Study Director — Centre for Rehabilitation Research
Locations (1):
- Hälsobro, Örebro, Örebro County, Sweden

REFERENCES:
- See also: Related Info — http://www.orebroll.se/sv/Forskning/Forskningsomraden/HFC1/personalHFC/Lars-Olov-Lundqvist/Kan-varken-tranas-bort/